CLINICAL TRIAL: NCT03153397
Title: Effect of Prebiotic Fiber- Enriched (scFOS) Enteral Feeding on the Microbiome in Neurological Injury Trauma Patients (PreFEED Microbiome Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00081414
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Enteral Nutrition; Brain Injuries, Traumatic; ICU Admission
Keywords: trauma; brain; neurological; injury; enteral; tube; feeding; nutrition
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Neurologic Manifestations | interventions — Osmolite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutraflora scFOS (Experimental): prebiotic fiber-containing formula (Nutraflora scFOS)
  Interventions: Other: Nutraflora scFOS
- Osmolite (Active Comparator): non-prebiotic fiber containing formula (Osmolite)
  Interventions: Other: Osmolite

INTERVENTIONS:
Other: Nutraflora scFOS — prebiotic fiber (Nutraflora scFOS via Vital AF)
  Arms: Nutraflora scFOS
Other: Osmolite — non-prebiotic fiber containing formula (Osmolite)
  Arms: Osmolite

SUMMARY:
This study plans to learn more about the impact of enteral nutrition on bacteria in critically ill trauma patients with brain injury. Specifically, it seeks to understand the effect that a prebiotic containing enteral feeding formula (Nutraflora scFOS in Vital AF) has on the gut, oral, and skin bacteria. A prebiotic is a special form of dietary fiber that acts as a fertilizer for good bacteria. The prebiotic Nutraflora scFOS has been cleared by the U.S. Food and Drug Administration and is not considered investigational as used in this study. Enteral feeding is a way to give nutrition to critically ill people who are unable to eat.

ELIGIBILITY:
Inclusion Criteria:

1. Adult major neurological injury trauma patients between 18-70 years of age who have been admitted directly to trauma ICU following major trauma
2. Expected length of mechanical ventilation > 48 hours (as judged by admitting clinician)
3. Expected length of ICU stay > 3 days (as judged by admitting clinician)
4. Expected to survive > 48 hours (as judged by admitting clinician)
5. Requiring enteral nutrition at any time in Intensive Care Unit (ICU) stay
6. Chronic illnesses must be under control (as determined by the Principal Investigator).

Exclusion Criteria:

1. Previous hospitalization within one month prior to ICU admission (no hospital floor transfers to eliminate confounding effect of previous hospital therapy)
2. Use of prebiotic fiber containing enteral or oral formula or probiotic preparations within one week
3. Received antibiotics within the previous month
4. On steroids or immunosuppressants at time of admission
5. All transplant patients
6. Chronic inflammatory disease that requires steroids or other biologic therapy intervention (e.g.: RA, IBD that requires steroids or Humira)
7. Undergoing active chemotherapy/radiation treatment
8. Renal failure requiring dialysis
9. Liver cirrhosis class C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in microbiome | Baseline (within 48 hours of ICU admission), up to 10 days
  Stool samples
Overall microbiome composition sampling gut | Baseline (within 48 hours of ICU admission), up to 10 days
  Stool samples
Change in microbiome longitudinally | Baseline at Day 2, 4, 6, 8 and 10
  Tongue swab microbiome longitudinally
Changes in the microbiome on delivery of initial clinical outcomes in trauma patients | Baseline (within 48 hours of ICU admission), up to 10 days
  Stool samples

SECONDARY OUTCOMES:
Record length of mechanical ventilation | Up to 60 days
Length of ICU | Up to 60 days
Length of hospital stay | Up to 60 days
Mortality | Up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serbanescu MA, Wright MC, Elebasy M, Shi P, Arnold JW, Haines KL, White JR, Surana NK, Wischmeyer PE. Impact of fiber-containing enteral nutrition on microbial community dynamics in critically ill trauma patients: a pilot-randomized trial. BMC Med. 2025 Dec 29;23(1):706. doi: 10.1186/s12916-025-04511-2. PMID 41462238